CLINICAL TRIAL: NCT00261131
Title: Efficacy and Functional Outcomes of Botulinum Toxin A Injections to Hamstrings in Flexed Knee Gait in Cerebral Palsy: A Double-Blind, Randomized, Placebo-Controlled Trial
Brief Title: Efficacy and Functional Outcomes of Botulinum Toxin A Injections to Hamstrings in Flexed Knee Gait in Cerebral Palsy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Shriners Hospitals for Children (Other)
Collaborators: University of Virginia (Other); Washington University School of Medicine (Other)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 9199
Record Dates: First submitted 2005-11-30; First posted 2005-12-02 (Estimated); Last update posted 2009-02-05 (Estimated); Status verified 2009-02

CONDITIONS: Spastic Diplegic Cerebral Palsy
Keywords: cerebral palsy; spasticity; diplegia
MeSH Terms: conditions — Cerebral Palsy; Muscle Spasticity | interventions — Botulinum Toxins, Type A

INTERVENTIONS:
Drug: Botulinum Toxin A

SUMMARY:
The study proposes to determine if injections of BTX-A to the hamstring muscles result in measurable physiologic changes not observed with normal saline injections in children with spastic diplegic cerebral palsy who walk with a flexed-knee gait pattern.

DETAILED DESCRIPTION:
This study proposes to: (1) to determine if injections of BTX-A to the hamstring muscles result in measurable physiologic (body structure and body function) changes not observed with normal saline injections, in children with spastic diplegic CP who walk with a flexed-knee gait pattern; (2) to assess whether physiologic changes translate into functional (activity and participation) improvements; (3) to evaluate family's perception of change in function, activity, participation, and quality of life.

This study will demonstrate if BTX-A injected into overactive hamstring muscles of children with spastic cerebral palsy (CP) and a flexed-knee walking pattern has measurable effects across the spectrum of dimensions of disablement of the International Classification of Functioning, Disability, and Health (ICF). It is a multi-center, prospective, randomized, double-blind trial comparing results of injection of BTX- A and placebo saline in controls, into overactive hamstring muscles, using multiple outcomes measures. Temporal-spatial gait parameters, instrumented 3DGA kinematics, passive ROM, spasticity measurement with both Ashworth and Tardieu scales, muscle strength/control, Gross Motor Function Measurement (GMFM), Pediatric Outcomes Data Collection Instrument (PODCI), Gillette Functional Assessment Questionnaire (FAQ), 6-Minute Walk Test, and Goal Attainment Scale (GAS), assessing all ICF domains, will be collected at baseline and at 1 month, 3 months, and 6 months post-injection. Power analysis demonstrates the need to randomize 250 children (125 with BTX-A, 125 with saline), allowing for attrition. Nine participating hospitals will contribute patients.

ELIGIBILITY:
Inclusion Criteria:

1. Spastic cerebral palsy;
2. Bilateral lower extremity involvement;
3. Spasticity present in the hamstrings;
4. Flexed knee gait >15 degrees by observation (OGS);
5. Age between 3 and 18 years old; (
6. GMFCS Level I to Level IV; (
7. Able to walk a minimum of 4 complete steps without resting with and without braces/shoes a minimum of 3 times;
8. Able to follow simple commands;
9. Cooperative with physicians and therapist;
10. Able to tolerate application of equipment to the skin.

Exclusion Criteria:

1. Rhizotomy surgery within the last 1 year;
2. Lower extremity surgical procedures (soft tissue or bony) within the past 1 year;
3. Currently implanted and operating Intrathecal Baclofen Pump (oral baclofen OK);
4. Lower extremity BTX-A injections within the past 6 months;
5. Multilevel BTX-A injections;
6. Gait trainer reliance;
7. Serial casting 3 months prior to or during study protocol.

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 250 (Estimated)
Dates: Start 2006-03; Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
3DGA Kinematics
Passive Range of Motion
Spasticity Measurement with AShworth and Tardieu Scales
Muscle Strength and Control

SECONDARY OUTCOMES:
Gross Motor Function Measurement (GMFM)
Pediatric Outcomes Data Collection Instrument (PODCI)
Gillette Functional Assessment Questionnaire (GFAQ)
6-Minute Walk Test
Goal Attainment Scale (GAS)

CONTACTS AND LOCATIONS:
Overall Officials: Philip E. Gates, MD, Principal Investigator — Shriners Hospitals for Children